CLINICAL TRIAL: NCT00272493
Title: Improving Immune Response to Hepatitis B Vaccine in HIV-positive Subjects Using Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) as a Vaccine Adjuvant: A Phase II Open-Label Pilot Study
Brief Title: Safety and Effectiveness of an Adjuvant in Improving Immune Response to Hepatitis B Virus Vaccine in HIV Infected Individuals
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A5220; 10148 (Registry Identifier: DAIDS ES Registry ID); ACTG A5220
Record Dates: First submitted 2006-01-04; First posted 2006-01-06 (Estimated); Last update posted 2021-10-25 (Actual); Status verified 2012-05

CONDITIONS: HIV Infections
Keywords: Treatment Experienced; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Hepatitis B Vaccines

ARMS (2):
- A (Active Comparator): Arm A participants will receive 40 mcg of HBV vaccine at study entry, Week 4, and Week 12.
  Interventions: Biological: Hepatitis B virus vaccine
- B (Experimental): Arm B participants will receive 40 mcg of HBV vaccine and 250 mcg of GM-CSF at study entry, Week 4, and Week 12.
  Interventions: Biological: Hepatitis B virus vaccine with GM-CSF adjuvant

INTERVENTIONS:
Biological: Hepatitis B virus vaccine with GM-CSF adjuvant — Arm B participants will receive 40 mcg of HBV vaccine and 250 mcg of GM-CSF at study entry, Week 4, and Week 12.
  Arms: B
Biological: Hepatitis B virus vaccine — Arm A participants will receive 40 mcg of HBV vaccine at study entry, Week 4, and Week 12.
  Arms: A

SUMMARY:
Granulocyte-macrophage colony-stimulating factor (GM-CSF) is a naturally occurring substance that is made by the body in response to infection or inflammation, and greatly improves cellular immune responses. The purpose of this study is to evaluate the safety and effectiveness of GM-CSF as an adjuvant to improve the immune response to hepatitis B virus (HBV) vaccination in HIV infected individuals.

DETAILED DESCRIPTION:
Highly active antiretroviral therapy (HAART) has greatly improved the life of HIV infected individuals. Before the introduction of HAART, the impact of HBV infection and liver disease was less prominent due to the rapid progression to AIDS. However, with the use of HAART, liver disease has become a leading cause of death in HIV infected individuals; therefore, prevention of HBV infection is essential. Most HIV infected people respond poorly to HBV vaccines. GM-CSF is a cytokine produced primarily by activated T and B cells and has been used extensively as a hematopoietic growth factor. GM-CSF increases neutrophil count, improves antigen-presenting cell function, and is involved in the development and improvement of cellular immune responses. Past research has shown that GM-CSF improves the immune response to HBV vaccination in people with kidney disease. The purpose of this study is to evaluate the safety and effectiveness of GM-CSF as an adjuvant to improve the immune response to HBV vaccination in HIV infected individuals.

This study will last 60 weeks. Participants will be randomly assigned to 1 of 2 arms. Arm A participants will receive 40 mcg of HBV vaccine at study entry, Week 4, and Week 12. Arm B participants will receive 40 mcg of HBV vaccine and 250 mcg of GM-CSF at study entry, Week 4, and Week 12. Participants will be stratified by their screening HIV-1 viral load. After completing the vaccination series, study visits will occur at Weeks 16, 36, and 60. Blood collection, a physical exam, and liver function and hepatitis antibody tests will be completed at all study visits. Telephone follow-up by study staff will occur 48 to 96 hours post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* CD4 count of 200 cells/mm3 or more within 30 days prior to study entry
* HIV-1 RNA viral load value obtained within 30 days prior to study entry
* Received HAART for at least 8 weeks prior to study entry OR not on HAART within 8 weeks prior to study entry with no plans to start HAART during the study. Participants receiving HAART must be on stable therapy as defined by the protocol.
* Negative hepatitis B core total antibody (HBcAb total), qualitative hepatitis B surface antibody (HBsAb), and hepatitis B surface antigen (HBsAg) tests within 30 days prior to study entry
* Negative hepatitis C virus (HCV) antibody test, completed within 30 days prior to study entry
* Willing to use acceptable forms of contraception

Exclusion Criteria:

* HCV antibody or HCV RNA positive at any time prior to study entry
* Previously vaccinated against HBV
* Use of any systemic antineoplastic or immunomodulatory treatment, systemic corticosteroids, vaccines, interleukins, interferons, growth factors, or intravenous immune globulin within 30 days prior to study entry
* Known allergy or sensitivity to any component of the study drugs
* Active drug or alcohol dependence that would interfere with participation in the study
* Any mental illness that may interfere with the study
* Serious illness requiring systemic treatment or hospitalization. Participants who complete therapy or are clinically stable on therapy for at least 14 days prior to study entry are not excluded.
* Body weight less than 50 kg (110 lbs)
* Abnormal lab values
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Primary Completion 2007-11 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Quantitative hepatitis B surface antibody (HBsAb) | At Week 16
Occurrence of Grade 3 or higher adverse events (including hypersensitivity reaction) related to study regimens and HIV viral load increase greater than 1 log(10) | Throughout the study

SECONDARY OUTCOMES:
Quantitative HBsAb 24 and 48 weeks after completion of HBV vaccination series | At Weeks 36 and 60
HBsAb response, defined as titer greater than 10 mlU/ml at 4, 24, and 48 weeks after completion of HBV vaccination series | At Weeks 16, 36, and 60
Changes in HIV viral load from baseline | At Weeks 4, 16, and 60
Changes in white blood cell and absolute neutrophil count from baseline | At Weeks 4, 16, and 36
Occurrence of Grade 2 or higher adverse events | Throughout the study
Changes in CD4 count from baseline | At Weeks 4, 16, and 60

CONTACTS AND LOCATIONS:
Overall Officials: Judith A. Aberg, MD, Study Chair — New York University; Edgar (Turner) Overton, MD, Study Chair — AIDS Clinical Trials Unit, Washington University at St. Louis
Locations (11):
- United States (11):
  - Northwestern University CRS, Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Washington U CRS, St Louis, Missouri
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Univ. of Rochester ACTG CRS, Durham, North Carolina
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Case CRS, Cleveland, Ohio
  - MetroHealth CRS, Cleveland, Ohio
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
  - University of Washington AIDS CRS, Seattle, Washington

REFERENCES:
- [Background] Bica I, McGovern B, Dhar R, Stone D, McGowan K, Scheib R, Snydman DR. Increasing mortality due to end-stage liver disease in patients with human immunodeficiency virus infection. Clin Infect Dis. 2001 Feb 1;32(3):492-7. doi: 10.1086/318501. Epub 2001 Jan 23. PMID 11170959
- [Background] Laurence JC. Hepatitis A and B immunizations of individuals infected with human immunodeficiency virus. Am J Med. 2005 Oct;118 Suppl 10A:75S-83S. doi: 10.1016/j.amjmed.2005.07.024. PMID 16271546
- [Background] Sasaki Md, Foccacia R, de Messias-Reason IJ. Efficacy of granulocyte-macrophage colony-stimulating factor (GM-CSF) as a vaccine adjuvant for hepatitis B virus in patients with HIV infection. Vaccine. 2003 Nov 7;21(31):4545-9. doi: 10.1016/s0264-410x(03)00500-0. PMID 14575766
- [Background] Thio CL, Seaberg EC, Skolasky R Jr, Phair J, Visscher B, Munoz A, Thomas DL; Multicenter AIDS Cohort Study. HIV-1, hepatitis B virus, and risk of liver-related mortality in the Multicenter Cohort Study (MACS). Lancet. 2002 Dec 14;360(9349):1921-6. doi: 10.1016/s0140-6736(02)11913-1. PMID 12493258
- [Result] Overton ET, Kang M, Peters MG, Umbleja T, Alston-Smith BL, Bastow B, Demarco-Shaw D, Koziel MJ, Mong-Kryspin L, Sprenger HL, Yu JY, Aberg JA. Immune response to hepatitis B vaccine in HIV-infected subjects using granulocyte-macrophage colony-stimulating factor (GM-CSF) as a vaccine adjuvant: ACTG study 5220. Vaccine. 2010 Aug 2;28(34):5597-604. doi: 10.1016/j.vaccine.2010.06.030. Epub 2010 Jun 23. PMID 20600512
- [Derived] Anthony DD, Umbleja T, Aberg JA, Kang M, Medvik K, Lederman MM, Peters MG, Koziel MJ, Overton ET. Lower peripheral blood CD14+ monocyte frequency and higher CD34+ progenitor cell frequency are associated with HBV vaccine induced response in HIV infected individuals. Vaccine. 2011 Apr 27;29(19):3558-63. doi: 10.1016/j.vaccine.2011.02.092. Epub 2011 Mar 11. PMID 21397720